CLINICAL TRIAL: NCT05733247
Title: The Effect of 6 Week Adductor Exercise Programs on Adductor Muscle Function and Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dublin City University (Other)
Responsible Party: Principal Investigator, Enda Whyte, Assistant professor, Dublin City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022_ATT_EW_14
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Adductor Strain
Keywords: Hip adductor; Hip abductor; groin injuries; Copenhagen adductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copenhagen adductor exercise (Active Comparator): The modified Copenhagen adductor exercise consists of 6 levels through which the participant will progress when able to complete one level adequately (able to complete the exercise in the given timeframe with adequate control). The first 5 levels are isometric contractions progressing in difficulty with the 6th level including concentric and eccentric components.
  1. Participants perform a supported isometric adduction hold off a 30cm support in a short-lever side-lying position. The participants then raise their pelvis from the floor, keeping their lower knee on the ground for support and hold for 20 seconds, repeating it twelve times on each side.
  2. Participants progressed level 1 by lifting their supporting leg, bringing their knees together and holding position for 20 seconds, repeating it twelve times on each side.
  Interventions: Other: Copenhagen adductor exercise
- adduction and abduction partner exercise (Experimental): Participants are in a sitting position with their knees extended and hips abducted, supporting themselves with their hands behind their trunks, facing each other. For the adduction exercise, the participant will place his feet and lower leg on the outside of his partner's lower legs and feet. He will then adduct his hips, bringing his feet slowly together while his partner slowly resists this movement.
  For the abduction exercise, the participant will place his feet and lower legs on the inside of his partner's feet and lower legs. The participant will slowly abduct the hips while the partner resists this movement.
  Both exercises are performed over 6 seconds (a three second concentric and three second eccentric contraction) with as maximal effort.
  Interventions: Other: The adduction and abduction partner exercise

INTERVENTIONS:
Other: Copenhagen adductor exercise — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 -3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise.
  Arms: Copenhagen adductor exercise
Other: The adduction and abduction partner exercise — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 -3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise.
  Arms: adduction and abduction partner exercise

SUMMARY:
This research project will investigate the effects of two 6-week adductor (hip muscle) exercise programmes on adductor muscle function and performance.

Measures of adductor muscle strength and performance (jump height, hopping and sprint) and self reported hip and groin function using a questionnaire will be recorded pre and post a 6-week period. A group of footballers will be recruited and randomly allocated to an intervention or control group. Two different intervention groups will complete two different, six-week adductor exercise programmes in addition to their regular training programme. The exercise programmes will last 15 minutes (approximately) per session, with 3 sessions per week. The control group will continue their regular training programme.

DETAILED DESCRIPTION:
Participants will be recruited from the local university sports clubs. Club chairpersons will be asked to send an email to club players. Players interested in participating in the study will be asked to attend a meeting where the study will be explained to them. Those who were interested will then be assessed for inclusion and exclusion criteria.

Group allocation:

A four block randomization method will be used to allocate participants to the Copenhagen adductor exercise protocol or the adduction and abduction partner exercise protocol.

Interventions:

Copenhagen adductor exercise protocol or the adduction and abduction partner exercise.

Testing procedure:

The isometric strength of the participants' hip adductors and abductors will be recorded before and after the exercise intervention.

A 10 point visual analogue scale will be used to record the level of muscle soreness experienced after each training session.

ELIGIBILITY:
Inclusion Criteria:

* free from hip and groin injury in the 6 months prior to the study • currently competing in team sports at least three occasions per week

Exclusion Criteria:

* history of a hip or groin injury in the 3 months prior to the study
* a history of involvement in an adductor strengthening, injury prevention programme in the 3 months prior to the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-05-06 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
isometric hip adductor and abductor strength | Change from baseline after 6 weeks
  The maximum isometric hip abductor and adductor strength is assessed with the participant being tested was in supine position, with the test-leg placed at the end of the examination table, and the opposite leg slightly flexed. The dynamometer is placed 5 cm proximal to the proximal edge of the lateral mal¬leolus or 5 cm proximal to the proximal edge of the medial malleolus for hip abduction and adduction, respectively. The dynamometer is externally fix¬ated by the tester's hand/arm placed between the wall and the dynamometer. Participants are initially given two warm up trials of each test of the hip abductors and adductors at 50% and 100% of maximal voluntary isometric force (MVC), followed by three valid MVC trials at the rate of one trial every 60 s
Hop test function | Change from baseline after 6 weeks
  Single leg hop - the participant will hop as far forwards as possible. Triple hop for distance. Participants will be asked to hop forward three times in a row as far as possible.
  Crossover hop test. A 3 metre strip of tape will be place on the ground in front of the participants. Participants will be asked to stand on one foot with the tape to the outside of their stance foot. They will then be asked to hop forward three times in a row as far as possible while alternately crossing over the tape and then landing on the same foot, and holding this position for two seconds.
  Side hop test. Participants will be asked to jump from side to side as many times as possible in 30 seconds without touching the tape. The number of successful jumps will be recorded.

SECONDARY OUTCOMES:
Sprint performance | Change from baseline after 6 weeks
  all participants will perform three maximal 30 metre sprint tests with 4 minutes of recovery in between. Time elapsed will be recorded by timing gates placed at 0m, 5m, 15m, and 30m. Participants will start from a standing split position. The first timing gate will be triggered at initial toe off of the back leg. To account for the start of the sprint, a high speed 240Hz iPhone 6 camera and my sprint app will be used to adjust sprint times by calculating the time difference between toe off and the onset of initial movement. The camera will only be focussed on the participant's heel and there will be no images recorded that will identify a participant. Times will be recorded and mechanical sprint variables (maximal horizontal force production, maximal horizontal power output and maximal theoretical velocity) will be calculated using an Excel spreadsheet.The participants best time of the three attempts will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Enda Whyte, PhD, Principal Investigator — Dublin City University
Locations (1):
- Dublin City University, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No